CLINICAL TRIAL: NCT04249752
Title: New Biomarkers in Acute and Chronic Inflammatory Demyelinating Polyradiculoneuropathies
Brief Title: Biomarkers in Polyradiculoneuropathies
Acronym: BIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: CHU de la Timone, Marseille, France (Unknown); CHU Carémeau, Nîmes, France (Unknown); University Hospital, Bordeaux (Other); Centre hospitalier de Perpignan (Other); CH de Narbonne, France (Unknown); CH de Béziers France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0024
Record Dates: First submitted 2020-01-09; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Guillain-Barre Syndrome; CIDP
Keywords: chronic inflammatory demyelinating polyradiculoneuropathy; immunostaining; autoantibodies
MeSH Terms: conditions — Guillain-Barre Syndrome; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, lymphocyte, and cerebrospinal fluid,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 with GBS patients: GBS patients
- Group 2 with CIDP patients: with CIDP patients

SUMMARY:
The nodes of Ranvier contain ion channels that enable the rapid propagation of the nerve impulse. Cell adhesion molecules and glycolipids play an important role in the formation of the nodes of Ranvier. Antibodies against glycolipids are detected in half of patients with Guillain-Barré syndrome, an acute inflammatory neuropathy affecting peripheral nerve. The investigators found that antibodies target cell adhesion molecules at nodes of Ranvier in 10% of patients with chronic inflammatory demyelinating neuropathy (CIDP), another disabling neuromuscular disease affecting peripheral nerves. In the majority of patients with GBS or CIDP, the mechanisms responsible for the neuromuscular disorders are unknown. Our goals are to identify novel targets of antibodies in patients, this in order to find novel bio-markers and to better understand the physiopathology of inflammatory neuropathies. This work will help patient diagnosis and treatment orientation.

DETAILED DESCRIPTION:
Background: Inflammatory demyelinating polyradiculoneuropathies are rare disabling autoimmune diseases affecting the peripheral nervous system. These neuropathies can be acute, when signs and symptoms raise in less than 1 month (Guillain-Barré syndrome, GBS), or chronic, when deteriorations continue over more than 2 months from onset (CIDP). About half of GBS patients present with IgG1 or IgG3 anti-gangliosides antibodies. Gangliosides are glycolipidic structures mainly localized at the node and paranode areas. In CIDP patients, IgG4 auto-antibodies directed against nodal (Nfasc-186) or paranodal (Nfasc-155, CNTN1, Caspr-1) proteins are found in 5 to 10 %. In most GBS and CIDP patients, the antigenic target are unknown and clinical biomarkers are critically lacking to help diagnosis and treatment orientation. The aim of the present study is to identify new biomarkers in AIDP and CIDP patients.

Methods : The investigators conduct a national retrospective and prospective study to identify new antigenic targets in GBS and CIDP patients. Since 2015, the Institute for Neurosciences of Montpellier and the University Hospitals of Montpellier collect clinical, immulogical, electrophysiological, and histological data of GBS and CIDP patients. Each patient whose serum has already been collected gave written informed consent. GBS and CIDP are diagnosed according to the current criteria. Anti-gangliosides antibodies (by immunodot-blot) and anti-Nfasc155, -CNTN1, -Nfasc186, and -Caspr-1 antibodies (by ELISA and cell-binding assay) are assessed in GBS and CIDP patients, respectively. Among CIDP patients with monoclonal gammapathy, those presenting with anti-MAG antibodies, increasing VEGF, AL amyloidosis, and neurolymphomatosis are excluded. Patients' serum are also tested by immunohistochemical staining on wild-type and GalNacT -/- mouse sciatic nerve fibres.

Clinical and electrophysiological phenotypes are compared between patients with positive and negative immunostaining. Localization of the staining (i.e. node of Ranvier, paranodal region, and/or myelin sheath) as the subclass and isotype of the autoantibody are specified.

The search for a new antigenic target is performed in GBS and CIDP patients which are i) seronegatives for antiganglioside and anti-Nfasc155, -CNTN1, -Nfasc186, and -Caspr-1 antibodies, and presenting with ii) a postive immunostaining on wild-type and GalNacT-/- mouse sciatic nerve fibres. Then, serums of these selected patients are incubated with neuronal and glial cells in culture (spinal dorsal ganglia, motoneurons, Schwann cells, oligodendrocytes and neocortical neurons). In the case of positivity against cell culture, an immunoprecipitation is performed and the antigen/antibody complex is separated on SDS-PAGE 4-12% gel and electrophoretic bands are analyzed by mass spectrometry.

The aim of this study is to identify new antigenic targets in seronegative GBS and CIDP patients displaying immunoreactivity. The knowledge of these new targets may improve our diagnostic tools and could help to develop targeted therapies.

ELIGIBILITY:
Inclusion criteria:

* GBS or CIDP patients over 18 years old
* Signed informed consent
* With a positive immunostaining on wild-type and GalNacT-/- mouse sciatic nerve fibres.
* Subjects must be covered by public health insurance

Exclusion criteria:

- seropositive for anti-ganglioside, anti-MAG, and/or anti-Nfasc155, -CNTN1, -Nfasc186, and -Caspr-1 antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: GBS and CIDP patients according to the diagnostic criteria defined above.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between clinical features and immunoreactivity findings in GBS and CIDP patients | 24 months
  Correlation between the localization of the staining (i.e. node of Ranvier, paranodal region, and/or myelin sheath) and the axonal or demyelinating nature of the neuropathy (according to GBS and CIDP criteria).

SECONDARY OUTCOMES:
Screening and titration of antibodies against new antigenic targets in GBS and CIDP patients. | 5 years
  The serums of patients will be considered seropositives when optical density value is ≥ 0.1 in ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Taieb, MD, Study Director — UH MONTPELLIER
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC